CLINICAL TRIAL: NCT04303299
Title: A 6 Week Prospective, Open Label, Randomized, in Multicenter Study of, Oseltamivir Plus Hydroxychloroquine Versus Lopipinavir/ Ritonavir Plus Oseltamivir Versus Darunavir/ Ritonavir Plus Oseltamivir Plus Hydroxychloroquine in Mild COVID-19 AND Lopipinavir/ Ritonavir Plus Oseltamivir Versus Favipiravir Plus Lopipinavir / Ritonavir Versus Darunavir/ Ritonavir Plus Oseltamivir Plus Hydroxychloroquine Versus Favipiravir Plus Darunavir and Ritonavir Plus Hydroxychloroquine in Moderate to Critically Ill COVID-19
Brief Title: Fight COVID-19 Trial
Acronym: FIGHT-COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Principal Investigator, Dr Subsai Kongsaengdao, Associate Professor, Department of Medical Services Ministry of Public Health of Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-DMS-COVID19 study
Record Dates: First submitted 2020-02-24; First posted 2020-03-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: SARS-COV-2 Infections; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Masking Description: The study is described as 'open' unblinded, however all clinical, virological and laboratory data, as well as adverse events were reviewed by two independent physicians, and all radiological images were reviewed by two independent radiologists who were blinded to the treatment assignments.
  The study outcomes assessed blinded to randomized group ( PROBE design - prospective randomised open blinded evaluation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Oseltamivir plus Chloroquine in Mild COVID19 (Experimental): Oseltamivir 300mg ( or 4-6 mg/kg) per day plus Hydroxychloroquine 800 mg per day In mild COVID19
  Interventions: Drug: Oral
- Darunavir and Ritonavir plus oseltamivir (Experimental): Darunavir 400 mg every 8 hours Ritonavir 200 mg (or 2.5 mg/kg ) per day plus plus Oseltamivir 300mg ( or 4-6 mg/kg) per day plus Hydroxychloroquine 400mg per day in Mild COVID19
  Interventions: Drug: Oral
- Lopinavir and Ritonavir plus Oseltamivir in mild COVID19 (Experimental): Lopinavir 800 mg ( or 10 mg/kg ) per day and Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Oseltamivir 300 mg ( or 4-6 mg /kg ) per day In mild COVID19
  Interventions: Drug: Oral
- Lopinavir and Ritonavir Oseltamivir moderate to severe COVID19 (Experimental): Lopinavir 800 mg ( or 10 mg/kg ) per day and Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Oseltamivir 300 mg ( or 4-6 mg /kg ) per day In moderate to critically ill COVID19
  Interventions: Drug: Oral
- Favipiravir lopinavir /Ritonavir for mod. To severe (Experimental): Lopinavir 800 mg (or 10 mg/kg ) per day and Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Favipiravir 2400 mg, 2400 mg, and 1200 mg every 8 h on day 1, and a maintenance dose of 1200 mg twice a day in Mild COVID19 In moderate to critically ill COVID19
  Interventions: Drug: Oral
- Darunavir /ritonavir oseltamivir chloroquine mod-severe (Experimental): Darunavir 400 mg every 8 hours Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Oseltamivir 300 mg (or 4-6 mg /kg ) per day plus Hydroxychloroquine 400 mg per day In moderate to critically ill COVID19
  Interventions: Drug: Oral
- Darunavir /ritonavir favipiravir chloroquine mod-severe (Experimental): Darunavir 400 mg every 8 hours Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Favipiravir 2400 mg, 2400 mg, and 1200 mg every 8 h on day 1, and a maintenance dose of 1200 mg twice a day plus Hydroxychloroquine 400 mg per day In moderate to critically ill COVID19
  Interventions: Drug: Oral
- Conventional Qurantine (No Intervention): Patient who unwilling to treatment and willing to quarantine in mild COVID19

INTERVENTIONS:
Drug: Oral — Anti virus treatment
  Arms: Darunavir /ritonavir favipiravir chloroquine mod-severe; Darunavir /ritonavir oseltamivir chloroquine mod-severe; Darunavir and Ritonavir plus oseltamivir; Favipiravir lopinavir /Ritonavir for mod. To severe; Lopinavir and Ritonavir Oseltamivir moderate to severe COVID19; Lopinavir and Ritonavir plus Oseltamivir in mild COVID19; Oseltamivir plus Chloroquine in Mild COVID19

SUMMARY:
A 6-Week Prospective, Open label, Randomized, in Multicenter Study of, Oseltamivir 300mg per day plus Hydroxychloroquine 800 mg per day versus Combination of Lopipinavir 800mg (or 10 mg/kg ) per day and Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Oseltamivir 300 mg ( or 4-6 mg /kg ) per day versus Combination of Darunavir 400 mg every 8 hours plus ritonavir 200 mg (or 2.5 mg/kg ) per day plus Oseltamivir 300mg ( or 4-6 mg /kg ) per day plus Hydroxychloroquine 400 mg per day in mild COVID-19 and Combination of Lopipinavir 800 mg (or 10 mg/kg ) per day and Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Oseltamivir 300 mg ( or 4-6 mg /kg ) per day versus Favipiravir 2400 mg, 2400 mg, and 1200 mg every 8 h on day 1, and a maintenance dose of 1200 mg twice a day plus Lopipinavir 800 mg ( or 10 mg/kg ) per day and Ritonavir 200 mg ( or 2.5 mg/kg ) per day versus Combination of Darunavir 400 mg every 8 hours plus ritonavir 200 mg (or 2.5 mg/kg ) plus Oseltamivir 300 mg (or 4-6 mg /kg ) per day plus Hydroxychloroquine 400 mg per day versus Favipiravir 2400 mg, 2400 mg, and 1200 mg every 8 h on day 1, and a maintenance dose of 1200 mg twice a day plus Darunavir 400 mg every 8 hours Ritonavir 200 mg ( or 2.5 mg/kg ) per day plus Hydroxychloroquine 400 mg per day in moderate to critically illness in COVID-19

DETAILED DESCRIPTION:
Overall Study Design and Plan Various Combination of Protease inhibitors, Oseltamivir, Favipiravir, and Chloroquin for treatment of COVID-19. Non parametric and parametric statistical analysis will be analysed in the efficacy of treatment. For the pair-wise comparison, 2-sided p-value was used to ensure that the overall Type I error=0.05. Beta error 80%. Demographic and safety analyses were based on the summary of descriptive statistics.

Pre-randomization Phase The pre-randomization phase consisted of a screening period (0 to 1 day prior to randomization).

Screening Period (Day -1 to 0) At the screening visit and prior to performance of any study procedures, the investigators would explain the details of the study and the subject would have to sign on the written informed consent, exclusion criteria, and inclusion criteria Each subject who was willing to enrol into the study was asked about their medical history as well as their recent and current medications being taken. All enrolled subjects were asked to undertake an initial physical examination and had to satisfy the criteria for the inclusion /exclusion before being enrolled into the study.

All patients were asked to complete physical examination, CXR, CBC plt, proBNP, High sensitive C reactive protein and Laboratory blood (livers tests, haematology,) examinations, urine pregnancy test) were performed amount 5.5 mL for safety reasons. Nasopharyngeal swabs were collected to detect the ORF 1ab and E genes (sensitivity: 1000 copies per milliliter) by polymerase chain reactions. Will be performed The inclusion visit included the following examination and tests: - physical examination,- vital signs,- weight,- CBC laboratory test result,-Chest X ray or CT chest Blood for plasma cytokine assay -Pro BNP and High sensitive C reactive protein, D dimer Treatment period All patient will be treated with specific arm for 10-14 days or until negative for Nasopharyngeal swabs were collected to detect the ORF 1ab and E genes of SARS -CoV-2 for 3 consecutive tests every 24 -48 hours. ECG monitoring for prolonged QTcB in Hydroxychloroquine arm will be closed monitored The quarantine period will be performed for 7-14 days after swab negative All cases may be treated with Antibiotics as prophylaxis or specific treatment Other standard treatment will be allowed for investigator judgments. CXR nasoparyngeal swab will be performed every 1-2 days or up to investigator judgments Follow up Visits Patient will be check up CXR and CT scan, nasoparyngeal swab will be performed every 1-2 day until negative test and until 4-6 weeks or clinical complete recovery.

ELIGIBILITY:
Inclusion Criteria:

* The subject has to grant permission to enter into the study by signing and dating the informed consent form before completing any study-related procedure such as any assessment or evaluation not related to the normal medical care of the subject.
* Able to give written inform consent and retained one copy of the consent form
* Male or female subject, aged between 16 - 100 years old.
* Subject diagnosed to be COVID19
* Female subject in good health and sexually active was instructed by the investigator to avoid pregnancy during the study and to use condom or other contraceptive measure if necessary. The subject was required to have a negative urine pregnancy test before being eligible for the study. (At each of the subsequent visit, a urine pregnancy test was performed).
* Subject judged to be reliable for compliance for taking medication and capable of recording the effects of the medication and motivated in receiving benefits from the treatment.and compliance to quarantine procedure 7-14 days after treatment

Exclusion Criteria:

* The subject was pregnant or lactating.
* The subject was a female at risk of pregnancy during the study and not taking adequate precautions against pregnancy.
* The subject had a known hypersensitivity to any of the test materials or related compounds.
* The subject was unable or unwilling to comply fully with the protocol.
* Treatment with investigational drug (s) within 6 months before the screening visit.
* The subject had previously entered in this study.
* Patient who planned to schedule elective surgery during the study
* The used of other antiviral agents

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-28 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 eradication time | Up to 24 weeks
  Eradication of nasopharyngeal SARS-CoV-2

SECONDARY OUTCOMES:
Number of patient with Death | Up to 24 weeks
  Any death after treatment adjusted by initial severity in each arm
Number of patient with Recovery adjusted by initial severity in each arm | Up to 24 weeks
  Normal pulmonary function, normal O2 saturation after treatment Adjusted by initial severity in each arm
Number of day With ventilator dependent adjusted by initial severity in each arm | Up to 24 weeks
  Number of day with ventilator assistant
Number of patient developed Acute Respiratory Distress Syndrome After treatment | Up to 24 weeks
  Number of patient developed new ARDS

OTHER OUTCOMES:
Number of patient with Acute Respiratory Distress Syndrome Recovery | Up to 24 weeks
  Acute Respiratory Distress Syndrome Recovery rate
Time to recovery | Up to 24 Weeks
  The time to recovery was defined as the time between the first day of antiviral treatment or hospitalization to the day when there was no further requirement for antiviral medication or on-going medical care or the day of discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistant Professor Subsai Kongsaengdao, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Data references: Thai government data — https://ddc.moph.go.th
- Available data/document: News — https://world.kbs.co.kr/service/news_view.htm?lang=e&Seq_Code=151108
- Available data/document: Reference News — https://world.kbs.co.kr/service/news_view.htm?lang=e&Seq_Code=151108